CLINICAL TRIAL: NCT05484141
Title: The Effect of Blood Flow Restriction Applied to the Extensor Muscles on Muscle Architecture and Strength, Knee Pain, and Functions in Minor Patellar Instability
Brief Title: The Effect of Blood Flow Restriction Method in Patellar Instability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Begum Kara Kaya, Lecturer, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PFI
Record Dates: First submitted 2022-07-26; First posted 2022-08-02 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Patellar Abnormality
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Blood Flow Restriction (Experimental)
  Interventions: Other: Rehabilitation with blood blow restriction
- Without Blood Flow Restriction (Active Comparator)
  Interventions: Other: Rehabilitation without blood flow restriction

INTERVENTIONS:
Other: Rehabilitation with blood blow restriction — The rehabilitation program will be applied 2 days a week, for total of 8 weeks.
  Arms: With Blood Flow Restriction
Other: Rehabilitation without blood flow restriction — The rehabilitation program will be applied 2 days a week, for total of 8 weeks.
  Arms: Without Blood Flow Restriction

SUMMARY:
The blood flow restriction method, the effects of which have been frequently investigated in the literature in recent years, can produce muscle hypertrophy with low-intensity load and can be easily tolerated through to low mechanical stress, seems to be an exercise approach that can be used in the recovery of strength in cases with minor patellar instability and can contribute to the recovery of functional capacity without delay.

DETAILED DESCRIPTION:
Patellar instability is defined as disruption of normal movement of the patella in the trochlear groove, symptomatic, medial-lateral displacement. Patients with patellar instability may not be able to tolerate high-intensity quadriceps exercises in the early period of strengthening programs due to pain symptoms, and therefore strength recovery may be delayed. However, it is important to restore muscle strength, especially vastus medialis obliquus strength, as early as possible in patellar instability. The blood flow restriction method, the effects of which have been frequently investigated in the literature in recent years, can produce muscle hypertrophy with low-intensity load and can be easily tolerated through to low mechanical stress, seems to be an exercise approach that can be used in the recovery of strength in cases with minor patellar instability and can contribute to the recovery of functional capacity without delay.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-40 years,
* Volunteering to participate in the study,
* Having a complaint of anterior knee pain for at least 3 months,
* Having been diagnosed with unilateral minor patellar instability,
* Absence of any other ongoing clinical problems that interfere with exercise (will be questioned by the Physical Activity Readiness Questionnaire for All).

Exclusion Criteria:

* History of one or more traumatic-atraumatic patella dislocations,
* Evidence of osteoarthritis on radiological imaging (≥ Kellgren-Lawrence Stage 2)
* Having at least one of the contraindications preventing the application of blood flow restrictive exercises (Smoking, previous venous thromboembolism, risk of peripheral vascular disease (ankle-brachial index <0.9), coronary heart disease, hypertension, hemophilia, etc.),
* Previously diagnosed cardiovascular disease limiting effort capacity (Myocardial infarction, angina, exercise intolerance, etc.),
* Previously diagnosed neurological disorder or cognitive dysfunction (stroke, dementia, schizophrenia, etc.),
* Orthopedic lower extremity surgery in the last 1 year,
* Body mass index ≥ 30 kg/m2.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Muscle Architecture and Hypertrophy | 8 weeks
  A portable, diagnostic B-mode ultrasound device with a linear probe will be used to evaluate the quadriceps muscle architecture. Cross-sectional areas, muscle thicknesses, fascicle lengths, and pennation angles, the architectural parameters of both thigh muscles, will be assessed by ultrasound. All assessments will be calculated as millimeters.

SECONDARY OUTCOMES:
Assessment of Muscle Strength | 8 weeks
  The concentric and eccentric strength of the knee extensor muscle (quadriceps) and its antagonist (hamstring), will be measured using the isokinetic dynamometer.
Assessment of Pain | 8 weeks
  Visual Analogue Scale (VAS) will be used to evaluate the severity of pain in the knee of patients during activity, at rest, and at night. In the evaluation of pain intensity with VAS, the patient is asked to mark his pain above the 10-centimeter line defined as "0-no pain" and "10 unbearable pain" at both ends.
Evaluation of Functions | 8 weeks
  The Tampa Kinesiophobia Scale (TKS) will be used to evaluate kinesiophobia. The lower extremity functional capacity of the subjects will be evaluated with the 1-minute sit-to-stand test, and the knee functions will be evaluated with the Lysholm Knee Scoring Scale and the Kujala Patellofemoral Joint Evaluation Scale, which are patient-answered scales that are recommended to be used in cases with patellar instability. In addition, fatigue determination after each application will be made with the Borg CR-10 Perceived Fatigue Scale. Scales will be filled by the face-to-face evaluation method.
Evaluation of Satisfaction and Change | 8th week
  General satisfaction and the change in clinical status perceived by the participants will be evaluated with the 7 points Global Rating of Change Scale after the rehabilitation program. According to the scale, it is expressed as "-3: I am much worse, -2: I am worse, -1: I am a little worse, 0: No change, 1: I am a little better, 2: I am better, 3: I am much better".

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Zengin Alpözgen, PhD, Study Director — Istanbul University - Cerrahpasa

IPD SHARING:
Plan to Share IPD: No